CLINICAL TRIAL: NCT03174652
Title: Causes and Impact of Anemia on Pregnancy Outcome on the Thai-Myanmar Border: Retrospective Analysis
Brief Title: Anemia Pregnancy Outcome on the Thai-Myanmar Border
Acronym: AnPREG
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1703
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2017-08

CONDITIONS: Anemia Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The global burden of maternal morbidity and mortality attributable to anemia is staggering, and this is especially true in low-resource settings. A recent review suggests 42% of pregnant women have anemia worldwide (1993-2005) with the vast majority of anemic women (90%) residing in Africa or Asia1; and in Asia, anemia was the second highest cause of maternal mortality2. Anemia was diagnosed in almost one third to one half of women presenting to the Shoklo Malaria Research Unit (SMRU) clinics on the Thai-Myanmar border for antenatal care (ANC) in a 2008 survey3, and anemia at first antenatal visit was associated with a two-fold increase in maternal mortality in this population4. Studies have also shown an association between anemia and small for gestational age infants, preterm delivery, infant and childhood anemia and developmental delays5.

The anemia in pregnant women presenting to SMRU clinics is multifactorial, as hemoglobinopathies, Glucose-6-dehydrogenase (G6PD) deficiency, iron, folic acid and B12 deficiency, helminth infection, and malaria are all prevalent in this rural population. Though all of these pathologies can cause anemia, they require different and sometimes conflicting treatment and prevention strategies, interacting in a complex web of causes and effects. Iron supplementation is the mainstay of most anemia control programs, but some women with hemoglobinopathies suffer from potentially fatal iron overload6. Iron supplementation has also been associated with increased risk of malaria7. Some helminth infections are associated with increased rates of anemia and malaria, but others may be protective8. Malaria and G6PD deficiency have complex effects on one another, and some malaria treatments can cause acute and life-threatening hemolysis in G6PD deficient individuals9.

Given the high prevalence and diverse causes of anemia in this population, and its potentially dire effects on maternal and infant health and survival, SMRU implemented increased clinical testing for pregnant women in 2012 to inform clinical care at the individual level. Further analysis of these data is urgently needed to improve care on a population scale. We propose to review existing data from ANC records to determine the causes and effects of anemia in this population, and use this information to improve treatment and prevention guidelines. Results would be integrated rapidly into local practice with the potential to have profound impacts on maternal and child health in this region.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman voluntarily presented at SMRU antenatal clinics and at the first antenatal visit they were counselled about the types of tests that would be made available and that if they did not want to do them they could opt out and SMRU would still provide antenatal care, as for any other pregnant woman.

Exclusion Criteria:

* Women who chose to opt out of clinical sampling were excluded. Additionally, a very small number of women who were unstable at presentation to SMRU clinics were not sampled if sampling would have interfered with their clinical care.

However, since samples were generally clinically indicated to guide care in these patients, the majority did have testing done.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Data from approximately 15,548 new pregnant women enrolled to antenatal care from antenatal care (ANC) services of Shoklo Malaria Research Unit (SMRU) clinics during August 2012 to 31-Dec-2016.
Sampling Method: Non-Probability Sample
Enrollment: 13520 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Hematology | 1 year
  The contribution of thalassemia/other inherited red blood cell (IRBC) abnormalities to anemia in pregnant refugee and migrant Myanmar women attending antenatal clinics in a low resource setting.

SECONDARY OUTCOMES:
Hematology | 1 year
  The interaction between thalassemia/ other IRBC abnormalities and environmental (nutritional and infectious) causes of anemia
Serum ferritin | 1 year
  The pattern of iron stores (measured by serum ferritin) in pregnant women with thalassemia/ other IRBC abnormalities
The risk of maternal morbidities | 1 year
  The risk of maternal morbidities (especially gestational diabetes, preeclampsia, miscarriage) and/or infant morbidities (small for gestational age, stillbirth, anemia, predisposition to infection in the first year of life) in pregnancies with maternal thalassemia/other IRBC abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes